CLINICAL TRIAL: NCT00772642
Title: Profiling Immunological Parameters in the Cord Blood of Neonates Exposed to Plasmodium Falciparum in Utero
Brief Title: Immune Parameters in the Cord Blood of Newborns Exposed to Malaria in the Womb
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909004; 09-I-N004
Record Dates: First submitted 2008-10-11; First posted 2008-10-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-10

CONDITIONS: Malaria
Keywords: Cross-Sectional; Plasmodium Falciparum Malaria; Cord Blood; Immunology; Mali; Malaria
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study, conducted by the Malaria Research and Training Center at the University of Bamako, Mali, and the NIAID, will examine how exposure to the malaria parasite in the womb affects the developing immune system of newborns. Little is known about how such exposure in the womb may affect the immune system or alter the risk of malaria or responsiveness to vaccination after birth. A better understanding of this process may provide information useful for childhood vaccination strategies in areas where malaria is widespread.

Women 18 years of age and older who live in Bancoumana and are in their last trimester of pregnancy and in good health may be eligible for this study.

Participants have blood samples drawn from a finger stick and through a needle placed in a vein two times for this study: when they enroll in the study and again when they go to the Bancoumana Health Center to deliver their baby. After the baby and placenta are delivered, blood is collected from the umbilical cord and placenta.

...

DETAILED DESCRIPTION:
In malaria endemic areas the fetus is at risk for in utero exposure to Plasmodium falciparum or its soluble products. Little is known about how this exposure modulates the developing fetal immune system, or how this may alter the risk of malaria or responsiveness to vaccination after birth. A clearer understanding of this process may inform childhood vaccination strategies in malaria endemic areas. The objective of this cross-sectional exploratory study is to define the immune profile associated with in utero exposure to P. falciparum by analyzing cord blood samples collected at a site of high malaria transmission in Mali, and to compare this profile to that of U.S. cord blood samples. Pregnant women will be invited to participate in this study during the 3rd trimester of pregnancy. A finger stick blood draw will be collected from the mother at enrollment and peri-partum to determine if she is infected with P. falciparum. Cord blood and placental blood samples will be collected post-partum and processed to obtain mononuclear cells and serum. Cord blood can be obtained from the placenta after delivery without risk to mother or infant and will be used for research purposes only. Mononuclear cells will be analyzed by flow cytometry to characterize subsets of B, T and innate immune cells. Functional assays such as the B and T cell ELISPOT assay and measurements of cytokines in response to in vitro stimulation will also be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years
* Healthy female in 3rd trimester of pregnancy
* Resident of Bancoumana
* Willingness to allow cord and placental blood samples to be stored and used for future studies of the immune response to malaria
* Ability to give informed consent and willingness to comply with study requirements and procedures

EXCLUSION CRITERIA:

* Currently taking corticosteroids or other immunosuppressants
* Underlying heart disease, bleeding disorder, or other condition that in the judgment of the Principal Investigator (PI) could increase the risk to the volunteer
* Fever greater than or equal to 37.5 degree C or evidence of an acute infection
* Anemia (hemoglobin less than 9 g/dL)
* Participation in another clinical protocol that requires the administration of an experimental vaccine or experimental treatment.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-10-08; Study Completion 2010-09-10

CONTACTS AND LOCATIONS:
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Breman JG. The ears of the hippopotamus: manifestations, determinants, and estimates of the malaria burden. Am J Trop Med Hyg. 2001 Jan-Feb;64(1-2 Suppl):1-11. doi: 10.4269/ajtmh.2001.64.1. PMID 11425172
- [Background] Brustoski K, Kramer M, Moller U, Kremsner PG, Luty AJ. Neonatal and maternal immunological responses to conserved epitopes within the DBL-gamma3 chondroitin sulfate A-binding domain of Plasmodium falciparum erythrocyte membrane protein 1. Infect Immun. 2005 Dec;73(12):7988-95. doi: 10.1128/IAI.73.12.7988-7995.2005. PMID 16299291
- [Background] Desowitz RS. Prenatal immune priming in malaria: antigen-specific blastogenesis of cord blood lymphocytes from neonates born in a setting of holoendemic malaria. Ann Trop Med Parasitol. 1988 Apr;82(2):121-5. doi: 10.1080/00034983.1988.11812218. PMID 2460040